CLINICAL TRIAL: NCT07231341
Title: Insulin Resistance in Gestational Diabetes Mellitus
Acronym: IRIS
Status: Recruiting | Type: Observational
Sponsor: University of Aarhus (Other)
Collaborators: Aarhus University Hospital (Other)
Responsible Party: Principal Investigator, Ninna Lund Larsen, MD, PhD student, University of Aarhus
Other Study IDs: 1-10-72-350-21
Record Dates: First submitted 2025-09-22; First posted 2025-11-17 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Gestational Diabetes Mellitus (GDM)
Keywords: GDM; Gestational diabetes mellitus; CGM; Continuous glucose monitoring; Pregnancy; Diabetes in pregnancy
MeSH Terms: conditions — Diabetes, Gestational

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Weeks
Biospecimen Retention: Samples Without DNA — Plasma/serum retained.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pregnant women diagnosed with gestational diabetes mellitus: Continuous glucose monitoring for 14 days during pregnancy in women diagnosed with gestational diabetes mellitus. Delivery data are recorded, thus participants are followed up to 12 weeks.

SUMMARY:
This prospective cohort study investigates glycaemic variability, assessed by continuous glucose monitoring (CGM), in pregnant women with gestational diabetes mellitus (GDM) and its association with fetal growth and related maternal and neonatal outcomes. Participants will undergo 14 days of CGM during pregnancy to characterise individual glycaemic patterns. Clinical and paraclinical data, including fasting plasma glucose, HbA1c, lipid profile, organ markers of pregnancy-related medical conditions, maternal weight gain, and blood pressure will be collected at two study visits. Oral glucose tolerance test (OGTT) 2-hour values will be obtained at diagnosis. All participants will receive standard GDM care and routine obstetric follow-up for assessment of fetal growth and wellbeing. Birth weight, birth weight z-scores, and relevant neonatal outcomes will be recorded after delivery.

Statistical analyses will be performed using Stata statistical software (StataCorp LLC, College Station, TX, USA). Continuous and categorical variables will be summarised using appropriate descriptive statistics. Associations between maternal glycaemic variability and neonatal as well as other maternal metabolic outcomes will be explored using suitable statistical methods, with adjustment for relevant covariates. Exploratory analyses may include additional glycaemic variability metrics and lipid parameters to further characterise maternal metabolic patterns.

DETAILED DESCRIPTION:
The aim of this prospective cohort study is to investigate glycaemic variability, assessed by continuous glucose monitoring (CGM), in pregnant women with gestational diabetes mellitus (GDM), and its association with fetal growth and related maternal and neonatal outcomes.

Participants will undergo CGM for 14 consecutive days during pregnancy to characterise individual patterns of glycaemic variability. Relevant clinical and paraclinical parameters, including fasting plasma glucose, HbA1c, lipid profile (total cholesterol, HDL cholesterol, LDL cholesterol, and triglycerides), organ markers of pregnancy-related medical conditions (including liver and renal function parameters), maternal weight gain, and blood pressure will be recorded at both the commencement and after completion of the monitoring period. Oral glucose tolerance test (OGTT) 2-hour values will be retrieved from the diagnostic visit.

All participants will receive standard clinical care for GDM, including dietary counselling and routine obstetric follow-up for assessment of fetal growth and wellbeing. Following delivery, clinically relevant maternal and neonatal data, including birth weight, birth weight z-scores, and information on pregnancy or neonatal complications, will be obtained from electronic medical records.

Statistical analysis plan

Continuous variables will be assessed for distributional characteristics and summarised using appropriate descriptive statistics. Categorical variables will be presented as frequencies and percentages.

Associations between maternal glycaemic variability indices and study outcomes - including neonatal birth weight z-scores and other secondary maternal and neonatal parameters (e.g., 2-hour OGTT values, HbA1c, fasting glucose, and neonatal hypoglycaemia) will be explored using appropriate statistical methods according to data type and distribution. Multivariable models may be applied to adjust for relevant maternal and pregnancy-related covariates, including maternal age, pre-pregnancy BMI, gestational age at delivery, parity, HbA1c, and other relevant covariates where applicable.

Comparisons of glycaemic and metabolic parameters between relevant subgroups will be conducted using suitable statistical techniques selected based on data characteristics and study objectives. Categorical outcomes will be analysed using appropriate methods for comparison of proportions.

Additional glycaemic variability metrics (SD, MAGE, CONGA, and J-index) will be considered as pre-specified exploratory outcomes and may be analysed, contingent on data completeness and scientific relevance, to further characterise maternal glycaemic patterns. Exploratory analyses of associations between maternal glycaemic variability and lipid parameters (total, HDL, and LDL cholesterol, and triglycerides) may likewise be conducted on a non-primary, hypothesis-generating basis. Lipid measures may also be included as covariates in multivariable models evaluating neonatal outcomes.

All analyses will be two-tailed, and statistical significance will generally be inferred at p < 0.05. Statistical analyses will be performed using Stata statistical software (StataCorp LLC, College Station, TX, USA; current version at time of analysis).

ELIGIBILITY:
Inclusion Criteria:

* All singleton pregnant women with gestational diabetes mellitus (GDM) between gestational age (GA) 28+0 and 34+6 attending the obstetric outpatient clinic at Aarhus University Hospital, Aarhus, Denmark or Gødstrup Hospital, Herning, Denmark will be offered participation.

Exclusion Criteria:

* Pre-gestational diabetes
* Age < 18 years
* Multiple pregnancies
* Chronic disease that is not well-controlled and is expected to influence study outcomes (including inflammatory diseases such as rheumatologic, gastroenterological, etc.)
* Treatment with systemic corticosteroids
* Smoking
* Women who are unable to understand the oral and written patient information

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Stated in eligibility criteria. According to in- and exculsion criteria the study population will be singleton pregnant women > 18 years of age, with gestational diabetes mellitus (GDM) between gestational age (GA) 28+0 and 34+6, without poorly controlled chronic diseases who are non-smokers and not treated with systemic corticosteroids.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-09-22 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Birth weight z-scores | Recorded immediately after delivery.
  Calculated using reference standards adjusted for gestational age and sex. Unit of measure: z-score (SD units).

SECONDARY OUTCOMES:
Maternal glycaemic variability, Coefficient of Variation (CV) | Measurements will be commenced between gestational week 28+0 and 34+6.
  Coefficient of variation (%) of interstitial glucose derived from 14 consecutive days of continuous glucose monitoring (CGM).
Maternal Time in Range (TIR) | Measurements will be commenced between gestational week 28+0 and 34+6.
  Percentage of time with blood glucose levels within the pregnancy target range (3.9 - 7.0 mmol/l) during the 14-day CGM period.
Maternal Time Above Range (TAR) | Measurements will be commenced between gestational week 28+0 and 34+6.
  Percentage of time with blood glucose levels above the pregnancy target range (3.9 - 7.0 mmol/l) during the 14-day CGM period.
Maternal Time Below Range (TBR) | Measurements will be commenced between gestational week 28+0 and 34+6.
  Percentage of time with blood glucose levels below the pregnancy target range (3.9 - 7.0 mmol/l) during the 14-day CGM period.
2-hour oral glucose tolerance test (OGTT) | Measured at diagnosis of gestational diabetes mellitus.
  2-hour venous plasma glucose following a 75-g oral glucose tolerance test performed during routine GDM screening. Unit of measure: mmol/L.
HbA1c | Maternal HbA1c levels measured at first study visit (gestational week 28+0 to 34+6) and at the second study visit (gestational week 30+0 to birth).
  Maternal HbA1c levels (mmol/mol, IFCC).
Fasting blood glucose | Measured at first study visit (gestational week 28+0 to 34+6) and after completion of the measurement period, at the second study visit (gestational week 30+0 to birth).
  Fasting venous plasma glucose (mmol/L).
Neonatal hypoglycaemia | From birth to 24 hours of life.
  Neonatal blood glucose <2.5 mmol/l.
Birth weight | Immediately after delivery.
  Absolute neonatal birth weight measured after delivery (grams).

OTHER OUTCOMES:
Maternal glycaemic variability, Standard Deviation (SD) | Measurements will be commenced between gestational week 28+0 and 34+6.
  Standard deviation of interstitial glucose from continuous glucose monitoring (CGM) over 14 consecutive days. Unit of measure: mmol/L. Measurement tool: FreeStyle Libre Pro IQ.
Maternal glycaemic variability, Mean Amplitude of Glycaemic Excursions (MAGE) | Measurements will be commenced between gestational week 28+0 and 34+6.
  MAGE calculated from CGM profiles over 14 consecutive days using a standard algorithm. Unit of measure: mmol/L.
Maternal glycaemic variability, J-index | Measurements will be commenced between gestational week 28+0 and 34+6.
  J-index computed from mean glucose and SD over the 14-day CGM period, using the prespecified formula (J-index = 0.001 × (mean + SD)²). Unit of measure: mmol/L.
Maternal glycaemic variability, CONGA | Measurements will be commenced between gestational week 28+0 and 34+6.
  Continuous Overall Net Glycaemic Action (CONGA) calculated over the prespecified lag (e.g., CONGA-1 or CONGA-2) from 14-day CGM data. Unit of measure: mmol/L.
Maternal lipid profile (total, HDL, and LDL cholesterol) | Measured at first study visit (gestational week 28+0 to 34+6) and after completion of the measurement period (gestational week 30+0 to birth).
  Maternal total cholesterol, high-density lipoprotein (HDL) cholesterol, and low-density lipoprotein (LDL) cholesterol measured in maternal venous blood using standardized enzymatic colorimetric assays at an accredited clinical laboratory. Unit of measure: mmol/L.
Maternal triglycerides | Measured at first study visit (gestational week 28+0 to 34+6) and after completion of the measurement period (gestational week 30+0 to birth).
  Serum triglyceride concentration measured in maternal venous blood using a standardized enzymatic colorimetric assay at an accredited clinical laboratory.
  Unit of measure: mmol/L.

CONTACTS AND LOCATIONS:
Overall Officials: Ninna L Larsen, MD, Principal Investigator — University of Aarhus
Locations (2):
- Denmark (2):
  - Aarhus University Hospital, Aarhus
  - Gødstrup Hospital, Herning

IPD SHARING:
Plan to Share IPD: No